CLINICAL TRIAL: NCT06266091
Title: A Phase II, Randomized, Open-label, Controlled, Multicenter Study to Evaluate the Efficacy and Safety of M701 Combined With Systemic Therapy in Patients With Malignant Ascites Caused by Gastrointestinal or Ovarian Cancer.
Brief Title: Treat Malignant Ascites Caused by Gastrointestinal or Ovarian Cancer With M701 Bispecific Antibody
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M70102
Record Dates: First submitted 2024-01-23; First posted 2024-02-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Malignant Ascites
MeSH Terms: interventions — Paracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- M701 group (Experimental): M701 will be administered via intra-peritoneal infusion following sufficient drainage of malignant ascites. The treatment regimen consists of a leading dose of 50μg on Day 1, followed by three infusions of the full dose of 400 μg M701 on Days 4, 11, and 18. If well tolerated, patients will continue to receive M701 infusions every 2 weeks as maintenance treatment. Additionally, these patients will receive systemic therapy as determined by the investigator.
  Interventions: Drug: M701
- Control group (Active Comparator): Patients in the control group will undergo paracentesis on Day 1 and Day 18. If necessary, they may receive additional paracentesis during this period. Additionally, these patients will receive systemic therapy as determined by the investigator.
  Interventions: Drug: paracentesis

INTERVENTIONS:
Drug: M701 — Intra-peritoneal infusion of M701 combined with system therapy
  Arms: M701 group
Drug: paracentesis — paracentesis combined with system therapy
  Arms: Control group

SUMMARY:
A Phase II, Randomized, Open-label, Controlled, Multicenter Study to Evaluate the Efficacy and Safety of M701 in treating Patients with Malignant Ascites Caused by Gastrointestinal or Ovarian Cancer combined with Systemic Therapy.

DETAILED DESCRIPTION:
The phase II study is a controlled, open-label trial designed to assess the effectiveness and safety of M701 intra-peritoneal infusion for controlling malignant ascites in patients with gastrointestinal and ovarian cancer who are also receiving systemic therapy.

A total of 80 patients with malignant ascites caused by gastrointestinal or ovarian cancer will be randomly assigned to two treatment arms in a 1:1 ratio. These patients must have experienced disease progression or intolerance after receiving at least two lines of systemic therapy. Both treatment arms will receive the systemic therapy, but the test arm will additionally receive M701 intra-peritoneal infusion, while the control arm will undergo paracentesis only.

The primary endpoint of the study will be the puncture-free survival, which evaluates the efficacy of M701 in controlling malignant ascites. Secondary endpoints include the objective response rate (ORR) of malignant ascites, progression-free survival (PFS), overall survival (OS), quality of life (QOL), and safety profiles. The number of EpCAM-positive cells in the malignant ascites will be measured using flow cytometry before and after treatment with M701.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign the written informed consent form.
* Histologically or pathologically confirmed epithelial malignancies, including advanced gastric cancer or colorectal cancer that has failed at least two lines of treatment, or platinum-resistant advanced ovarian cancer, primary peritoneal carcinoma, or fallopian tube carcinoma.
* Clinical diagnosis of malignant ascites with a moderate or higher amount of ascites. Moderate or higher is defined as having a volume of ascites ≥1L based on CT assessment or actual drainage of ≥1L.
* The time interval between the most recent anti-tumor treatment and the first dose of M701 must meet the following criteria:

Intraperitoneal treatment: ≥2 weeks since the most recent intraperitoneal treatment.

* Adverse events (AEs) from previous treatments have recovered to grade ≤1 (excluding other AEs deemed by the investigator not to affect the safety of the study drug, such as hair loss).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2. Estimated survival time ≥8 weeks.
* Organ function levels must meet the following requirements:

Hematology: Absolute neutrophil count (ANC) ≥1.5 × 10^9/L, platelets ≥80 × 10^9/L, hemoglobin ≥8.5 g/dL, lymphocyte ratio (lymphocyte count/leukocyte count) ≥10% (without transfusion within 14 days).

Liver function: Total bilirubin ≤1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times ULN (AST and ALT ≤5 times ULN allowed in the presence of liver metastasis).

Serum albumin ≥28 g/L. Renal function: Serum creatinine ≤1.5 times ULN.

Exclusion Criteria:

* Patients who have previously received M701 or any antibody-based drugs targeting EpCAM and/or CD3 within the 4 months prior to the first dose.
* Patients with microsatellite instability-high (MSI-H)/deficient mismatch repair (dMMR) colorectal cancer who have not previously received immunotherapy.
* Patients who have undergone major surgery within the 4 weeks prior to the first dose.
* Patients with extensive liver metastases (tumor volume occupying approximately >70% of total liver volume).
* Active infections requiring intravenous antibiotics within 14 days before the first dose.
* Severe diarrhea (CTCAE grade ≥2).
* Severe respiratory distress requiring oxygen therapy.
* Active autoimmune diseases, except for the following conditions that are allowed for screening: type 1 diabetes, controlled hypothyroidism with replacement therapy only, skin diseases that do not require systemic treatment。
* Other severe medical conditions that may limit the patient's participation in the trial。
* Impaired cardiac function with New York Heart Association (NYHA) class 3 or 4.
* Occurrence of complete intestinal obstruction within 30 days before the first dose, or diagnosis of incomplete intestinal obstruction deemed unsuitable for participation in the trial based on symptoms and signs as determined by the investigator.
* Inability to adequately drain ascites due to objective reasons (including loculated ascites).
* Confirmed portal vein obstruction.
* History of immunodeficiency, including positive HIV test.
* Active hepatitis B virus infection, active hepatitis C virus infection, active syphilis, or positive HIV antibody.
* Pregnant or lactating women.
* Patients with fertility requirements during or within 6 months after treatment.
* Known history of neurological or psychiatric disorders deemed by the investigator to affect cognitive function or compliance, including unstable epilepsy, dementia, schizophrenia, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Puncture-free survival, PuFS | From the time of 4th dosing (Day 18) to the next puncture/drainage or death (up to 6 months)
  The time to the next puncture/drainage or death

SECONDARY OUTCOMES:
objective response rate (ORR) of malignant ascites | From the time of 4th dosing (Day 18) to the next puncture/drainage or death (up to 180 days)re/drainage or death (up to 6 months)
  The change of precentage of malignant ascites volume from the baseline by the image evaluation
Progression-free Survival, PFS | From the time of first dosing (Day 1) until disease progression or toxicity intolerance or death (up to 6 months).
  The time to disease progression assessed by the imaging evaluation or toxicity or death
Overall survival, OS | From the time of first dosing (Day 1) until death (up to 6 months).
  The time to death
Quality of Life, QoL | From the time of first dosing (Day 1) until the EOT (up to 6 months).
  Using the QLQ-C30 Scale to score the quality of life at every visit, which includes 3 parts: global health status(2-14, higher is better), funtional status(16-64, lower is better), symptom scale(12-48, lower is better),
Safety profiles | From the time of first dosing (Day 1) until one month after the EOT (up to 6 months).
  frequency, relationship and seriousness of adverse events
Positive rate of ADA and Nab in serum | From the time of first dosing (Day 1) until the EOT (up to 6 months).
  The positive rate of Anti-Drug Antibody (ADA) and Neutralizing antibody (Nab) in the serum during the study
The EpCAM expression in ascites | From the time of first dosing (Day 1) until the EOT (up to 6 months).
  Measure the count of EpCAM postive cells in the ascites before and after M701 treatment
Trough serum concentration (Ctrough) | 6 months (anticipated)
  The lowest concentration of M701 in the serum in one treatment cycle
Peak serum concentration (Cmax) | 6 months (anticipated)
  The highest concentration of M701 in the serum in one treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, MD, Principal Investigator — The First Medical Center of Chinese PLA General Hospital
Locations (1):
- The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No